CLINICAL TRIAL: NCT00148512
Title: A Randomized, Double-blind, Placebo-controlled, Five Parallel Groups Efficacy and Safety Exploratory Study of NS 2330 (0.125 mg, 0.25 mg, 0.5 mg and 1.0 mg) Administered Orally Once Daily Over 14 Weeks in Levodopa Treated Parkinson Patients With Motor Fluctuations (Study for Proof of Concept in ADVAnced Parkinson Disease of NS 2330 / ADVANS)
Brief Title: A Randomized, Double-blind, Placebo-controlled, Five Parallel Groups Efficacy and Safety Study of NS 2330 (Tesofensine) (0.125 mg, 0.25 mg, 0.5 mg and 1.0 mg) Administered Orally Once Daily Over 14 Weeks in Levodopa Treated Parkinson Patients With Motor Fluctuations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1198.101
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Tesofensine

INTERVENTIONS:
Drug: 1. Tesofensine (NS 2330)

SUMMARY:
The primary objective of this exploratory study is to investigate the efficacy and safety of tesofensine in daily doses (from 0.125 mg to 1.0 mg) in comparison to placebo, over a 14-week treatment period in levodopa treated Parkinson patients with motor fluctuations.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, five parallel groups efficacy and safety exploratory of tesofensine versus placebo in levodopa treated Parkinson patients with motor fluctuations.

Patients will be treated either with one of the 4 doses of tesofensine (0.125mg, 0.25mg, 0.50 mg or 1.0 mg) or with placebo, once daily, over 14 weeks.

The two co-primary efficacy endpoints are the change in off-time and the change in the Unified Parkinson Disease Rating Scale (UPDRS) II+III total score

Study Hypothesis:

The null hypothesis is that there is no difference between placebo and tesofensine.

The alternative hypothesis is that treatment with tesofensine is superior to treatment with placebo.

Comparison(s):

For the primary comparison between tesofensine and placebo, change in percentage off-time during waking hours will be based on reports from patient's diary (completed at day -3 and day-2 prior to the study visits) and change in the UPDRS II+III will be based on UPDRS II averaged for on and off periods and UPDRS III evaluated at on periods during the study visits.

ELIGIBILITY:
Main inclusion criteria:

* Male or female patient with idiopathic Parkinson Disease (PD) diagnosed for at least 2 years.
* Patient aged 40 years or over at time of diagnosis of PD and not older than 80 years at screening visit.
* Modified Hoehn and Yahr stage of II to III at "on" time.
* Treatment with Levodopa at an optimised dose, 4 to 8 times per day, this dose being stable for at least 4 weeks prior to screening visit.
* Motor fluctuations, with 2.0 to 6.0 cumulative hours of "off" time every day during waking hours, documented from patient's diary completed for 2 consecutive days before baseline visit.

Main exclusion criteria:

* Neuropsychiatric exclusions: Non-idiopathic PD, dementia (Mini Mental State Exam <26), history of psychosis, history or current Axis I or Axis II mental disorder according to DSM-IV, etc
* Other medical exclusions, like ECG abnormalities, hypotension and/or symptomatic orthostatic hypotension, some abnormal laboratory parameters (e.g. severe renal impairment), etc
* Pharmacological exclusions, e.g. selegiline within 8 weeks prior to screening visit, regular use of anti-depressant drugs, any medication with central dopaminergic antagonist activity, etc

Ages: 42 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2003-03; Primary Completion 2005-02 (Actual); Study Completion 2005-02

PRIMARY OUTCOMES:
UPDRS parts II (averaged "on" and "off") | 14 weeks
"Off" time during waking hours | 14 weeks

SECONDARY OUTCOMES:
Percent on time without dyskinesia, or with non troublesome dyskinesia, or both, or with troublesome dyskinesia | 14 weeks
Unified Parkinson's Disease Rating Scale (UPDRS) I to IV sub-scores | 14 weeks
Clinical Global Impressions (CGI) Improvement and Severity | 14 weeks
Auditory Verbal Learning test (AVLT) | 14 weeks
Modified Schwab and England Disability scale | 14 weeks
Snaith-Hamilton Pleasure Scale (SHAPS) | 14 weeks
Percentage of patients with at least a 20%-improvement in percent "off" time during waking hours | 14 weeks
Percentage of patients with at least a 20% or a 30%-improvement in UPDRS parts II+III total score | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BI France S.A.S.
Locations (47):
- Austria (6):
  - Krankenhaus d. Barmherzigen Brüder Graz-Eggenberg, Graz
  - Univ.-Klinik für Neurologie, Graz
  - Univ.-Klinik für Neurologie, Innsbruck
  - Landesnervenklinik Wagner Jauregg Linz, Linz
  - AKH der Stadt Linz, Linz
  - Landesklinikum St. Pölten, Sankt Pölten
- France (10):
  - Hôpital du Pays d'Aix, Aix-en-Provence
  - Hôpital Pierre Wertheimer, Bron
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Roger Salengro, Lille
  - Hôpital de la Timone, Marseille
  - Service de Neurologie, Paris
  - Hôpital du Haut-Levèque, Pessac
  - Centre Hospitalier Universitaire JB Miletrie, Poitiers
  - Hôpital Guillaume et René Laennec, Saint-Herblain
  - Hôpital Purpan, Toulouse
- Germany (13):
  - Universitätsklinikum der Humboldt-Universität, Berlin
  - Boehringer Ingelheim Investigational Site, Berlin
  - St. Josef-Hospital, Bochum
  - Boehringer Ingelheim Investigational Site, Gera
  - Boehringer Ingelheim Investigational Site, Herborn
  - Paracelsus-Elena-Klinik, Kassel
  - Christian Albrechts Universität zu Kiel, Kiel
  - Universität Leipzig, Leipzig
  - Klinik für Neurologie, Marburg
  - Klinikum Großhadern der L.M.-Universität, München
  - Universitätsklinik Rostock, Rostock
  - Universitätsklinikum Ulm, Ulm
  - Deutsche Klinik für Diagnostik GmbH, Wiesbaden
- Netherlands (5):
  - Locatie Willem-Alexander, 's-Hertogenbosch
  - Boehringer Ingelheim Investigational Site, Breda
  - Martini ziekenhuis, Groningen
  - Maasland Ziekenhuis, Sittard
  - Boehringer Ingelheim Investigational Site, Utrecht
- Spain (6):
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Clinic i Provincial de BCN, Barcelona
  - Hospital de la Sta. Creu i Sant Pau, Barcelona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Clínico niversitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Clínico Universitario Vírgen de la Macarena, Seville
- United Kingdom (7):
  - City Hospital, Birmingham
  - Neurology Department, Blackburn
  - Neurology Department, Glasgow
  - Walton Centre for Neurology, Liverpool
  - Regional Neurosciences Centre, Newcastle upon Tyne
  - Neurology Research, Stoke-on-Trent
  - Neurology Department, Swansea

REFERENCES:
- [Derived] Rascol O, Poewe W, Lees A, Aristin M, Salin L, Juhel N, Waldhauser L, Schindler T; ADVANS Study Group. Tesofensine (NS 2330), a monoamine reuptake inhibitor, in patients with advanced Parkinson disease and motor fluctuations: the ADVANS Study. Arch Neurol. 2008 May;65(5):577-83. doi: 10.1001/archneur.65.5.577. PMID 18474731